CLINICAL TRIAL: NCT00664417
Title: Safety and Immunogenicity of Different Formulations of an Intramuscular A/H5N1 Inactivated, Split Virion Influenza Adjuvanted Vaccine in Healthy Adults
Brief Title: Study of Different Formulations of an Intramuscular A/H5N1 Inactivated, Split Virion Influenza Adjuvanted Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FUF04
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Influenza; Orthomyxoviridae Infections
Keywords: Influenza; A/H5N1; Orthomyxoviridae Infections; Influenza Pandemics
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 1 (Experimental)
  Interventions: Biological: Monovalent subvirion H5N1 influenza vaccine
- 2 (Experimental)
  Interventions: Biological: Monovalent subvirion H5N1 influenza vaccine
- 3 (Experimental)
  Interventions: Biological: Monovalent subvirion H5N1 influenza vaccine
- 4 (Experimental)
  Interventions: Biological: Monovalent subvirion H5N1 influenza vaccine
- 5 (Experimental)
  Interventions: Biological: Monovalent subvirion H5N1 influenza vaccine
- 6 (Experimental)
  Interventions: Biological: Monovalent subvirion H5N1 influenza vaccine
- 7 (Active Comparator)
  Interventions: Biological: Monovalent subvirion H5N1 influenza vaccine
- 8 (Active Comparator)
  Interventions: Biological: Monovalent subvirion H5N1 influenza vaccine
- 9 (Placebo Comparator)
  Interventions: Biological: Physiological saline

INTERVENTIONS:
Biological: Monovalent subvirion H5N1 influenza vaccine — 0.5 mL, IM, 2 injections, Formulation 1
  Arms: 1
Biological: Monovalent subvirion H5N1 influenza vaccine — 0.5 mL, IM, 2 injections, Formulation 2
  Arms: 2
Biological: Monovalent subvirion H5N1 influenza vaccine — 0.5 mL, IM, 2 injections, Formulation 3
  Arms: 3
Biological: Monovalent subvirion H5N1 influenza vaccine — 0.5 mL, IM, 2 injections, Formulation 4
  Arms: 4
Biological: Monovalent subvirion H5N1 influenza vaccine — 0.5 mL, IM, 2 injections, Formulation 5
  Arms: 5
Biological: Monovalent subvirion H5N1 influenza vaccine — 0.5 mL, IM, 2 injections, Formulation 6
  Arms: 6
Biological: Monovalent subvirion H5N1 influenza vaccine — 0.5 mL, IM, 2 injections, Comparator 1
  Arms: 7
Biological: Monovalent subvirion H5N1 influenza vaccine — 0.5 mL, IM, 2 injections, Comparator 2
  Arms: 8
Biological: Physiological saline — 0.5 mL, IM, 2 injections
  Arms: 9

SUMMARY:
Following the licensure of sanofi pasteur's 90 µg rgA/Vietnam/1203/2004 pandemic influenza vaccine, efforts to develop a lower antigen dose formulation with improved immunogenicity using adjuvants were initiated. The present study is part of this endeavor. It is primarily a formulation/dose-finding study with a secondary aim at generating safety and immunogenicity data for the final formulation for the development of a pre-pandemic vaccine.

DETAILED DESCRIPTION:
This is a Phase I, observer-blinded, randomized, controlled multicenter, dose-finding study in adult subjects. All vaccines will be administered as a two-dose schedule in (H5N1) immunologically-naïve adults. Immunogenicity and safety will be evaluated after each injection.

ELIGIBILITY:
Inclusion Criteria :

* Healthy adult aged 18 to 40 years on the day of inclusion.
* Provides signed informed consent prior to study procedures.
* Able to attend all scheduled visits and comply with all trial procedures.
* For a woman of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to the first vaccination, until at least 4 weeks after last vaccination.

Exclusion Criteria :

* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the standard-dose Fluzone® vaccine or to a vaccine containing any of the same substances
* For a woman of child-bearing potential, known pregnancy or positive serum/urine pregnancy test
* Breast feeding woman
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the (first) trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, oral, parenteral, or inhaled steroids
* Has an acute or chronic medical illness or any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or would interfere with the evaluation of responses or render the subject unable to meet the requirements of the protocol
* Known or suspected current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* History of receipt of blood or immunoglobulin or other blood-derived products within the 3 months prior to enrollment in this study that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination
* Planned receipt of any vaccine in the 4 weeks preceding or following any trial vaccination
* Known Human Immunodeficiency Virus (HIV), Hepatitis B surface antigen, or Hepatitis C seropositivity
* Personal or family history of Guillain-Barré Syndrome
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination
* Active neoplastic disease or a history of any hematologic malignancy
* Previous participation in a pandemic flu trial
* History of H5N1 infection or exposure to presumed/confirmed H5N1 human/animal cases
* Known seizure/epilepsy history and/or taking anti-seizure medication
* Receipt of psychiatric drugs. Subjects receiving a single antidepressant drug and stable for at least 3 months prior to enrollment, without decompensating symptoms will be allowed to enroll in the study.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 375 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety after primary administration of A/H1N1 vaccine | 6 months post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur, Inc.
Locations (5):
- United States (5):
  - San Diego, California
  - South Miami, Florida
  - Springfield, Missouri
  - Cincinnati, Ohio
  - Knoxville, Tennessee

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com